CLINICAL TRIAL: NCT00006088
Title: A Phase I Absolute Bioavailability Study of Oral NAVELBINE (Vinorelbine Tartrate) in Patients With Solid Tumors
Brief Title: Vinorelbine in Treating Patients With Metastatic or Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068080; MCC-11982; GW-VIN10003; NCI-G00-1826
Record Dates: First submitted 2000-08-03; First posted 2004-06-22 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2000-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Vinorelbine

INTERVENTIONS:
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase I trial to compare the effectiveness of two different regimens of vinorelbine in treating patients who have metastatic or advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the pharmacokinetic profiles of vinorelbine administered intravenously on day 1 and orally on day 8 vs the reverse order in patients with metastatic or advanced solid tumors. II. Determine the intersubject variability in the pharmacokinetics of oral vinorelbine. III. Compare the safety profiles of oral vs intravenous vinorelbine in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive vinorelbine IV over 20 minutes on day 1 and oral vinorelbine on day 8. Arm II: Patients receive oral vinorelbine on day 1 and vinorelbine IV over 20 minutes on day 8. Treatment continues in both arms in the absence of unacceptable toxicity or disease progression. Patients are followed for 28 days.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or advanced solid tumor that will potentially benefit from single agent vinorelbine No known CNS metastases unless successfully treated with excision or radiotherapy and stable for at least 6 months prior to study

PATIENT CHARACTERISTICS: Age: 18-75 Performance status: Not specified Life expectancy: Greater than 3 months Hematopoietic: Hemoglobin at least 9 g/dL (at least 3 weeks since last transfusion) Platelet count at least 75,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Transaminases no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN No unstable or uncontrolled hypercalcemia Cardiovascular: No venous access problems that would preclude blood sampling No symptomatic class II-IV congestive heart failure No significant ventricular arrhythmia requiring drug control No myocardial infarction within the past 6 months No uncontrolled cardiac disease or unstable angina No recurrent thromboembolic events No unstable or uncontrolled arterial hypertension Pulmonary: No history of recurrent aspiration pneumonitis or aspiration pneumonia No severe respiratory insufficiency, defined by oxygen partial pressure less than 60 mm Hg on room air and requirement for chronic oxygen therapy Gastrointestinal: See Surgery No active gastrointestinal disease or disorder that alters gastrointestinal motility or absorption No lack of integrity of the gastrointestinal tract No unstable or uncontrolled diarrhea or peptic ulcer disease Other: Able to receive IV and oral regimens Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for at least 2 weeks before, during, and for at least 9 days after study No preexisting peripheral neuropathy greater than grade 1 No active infection within the past 2 weeks No fever (temperature at least 37.5 degrees C) or other symptoms of possible infection within 10 days after completing antimicrobial treatment No psychological, familial, or sociological condition that would preclude study No unstable or uncontrolled preexisting medical condition (e.g., diabetes, alcohol withdrawal)

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior packed red blood cell transfusion At least 1 week since prior platelet transfusion or hematopoietic growth factors No concurrent growth factors earlier than 24 hours after study drug Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered No other concurrent antineoplastic agents Endocrine therapy: At least 3 weeks since prior hormonal therapy and recovered Concurrent megestrol allowed No other concurrent hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Prior or concurrent palliative radiotherapy to peripheral bone lesion, spinal cord compression, or imminent fracture allowed only if less than 10% of bone marrow involved Surgery: No prior significant surgical resection of the stomach or small bowel At least 2 weeks since prior surgery Other: No other concurrent experimental or anticancer drugs or devices At least 1 week since prior products or drugs known to induce or inhibit the enzymatic activity of vinorelbine (e.g., antihistamines, phenobarbital, meprobamate, some antiepileptics, or grapefruit juice) No concurrent products or drugs known to induce or inhibit the enzymatic activity of vinorelbine No concurrent opiates or laxatives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Sullivan, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States